CLINICAL TRIAL: NCT02337881
Title: Combined Nifedipine and Sildenafil Citrate Versus Nifedipine Alone in Acute Tocolysis of Preterm Labor: A Randomized Clinical Trial
Brief Title: Management of Acute Preterm Labor: Nifedipen Alone or Combined With Cildenafil Citrate
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al Hayat National Hospital (Other)
Collaborators: Menoufia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ob/gyn 2
Record Dates: First submitted 2014-12-30; First posted 2015-01-14 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Labor Preterm Requiring Hospitalization
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nifedipen and sildenafil (Active Comparator): The protocol for nifedipen in our units consists of 20 mg orally stat, followed by 10 mg orally every 6-8 hours, at the same time sildenafil citrate will be administered vaginally in a dose of 25mg at 8 hourly intervals and both medications will be continued for 48-72 hours as indicated.
  Interventions: Drug: nifedipen; Drug: Sildenafil
- nifedipen only (Active Comparator): nifedipine alone in the same regimen and duration described before.
  Interventions: Drug: nifedipen

INTERVENTIONS:
Drug: nifedipen — The protocol for nifedipen in our units consists of 20 mg orally stat, followed by 10 mg orally every 6-8 hours for 48 to 72 hours as needed
  Other Names: inhibiting acute preterm labor
Drug: Sildenafil — sildenafil citrate will be administered vaginally in a dose of 25mg at 8 hourly intervals and both medications will be continued for 48-72 hours as indicated.
  Other Names: inhibiting acute preterm labor
  Arms: nifedipen and sildenafil

SUMMARY:
The aim of this study is to assess whether or not the emergency tocolytic effect of combined nifedipine and sildenafil citrate will have a superior effect over nifedipine alone in terms of inhibiting eminent preterm labor and improving perinatal outcomes.

DETAILED DESCRIPTION:
Women will be randomly assigned into two study groups using a computerized random number table generator in order to get the trial sequence which will be hidden in sealed numbered opaque envelopes. Each envelope contains a single element (assignment) of the trial sequence. The statistician generated the random allocation sequence, and the investigators enrolled the participants.

Each patient will undergo an ultrasound examination prior to randomization to confirm GA, rule out major fetal anomalies and to determine cervical measurements. Dexamethasone in a total dose of 24 mg will be administered to all patients if not given in a previous admission.

Eligible women are then randomly assigned into two study groups:

Group I: (combined nifedipine and sildenafil citrate) The protocol for nifedipen in our units consists of 20 mg orally stat, followed by 10 mg orally every 6-8 hours, at the same time sildenafil citrate will be administered vaginally in a dose of 25mg at 8 hourly intervals and both medications will be continued for 48-72 hours as indicated.

Group II: (nifedipine alone) will receive therapy by nifedipine alone in the same regimen and duration described before.

During therapy, maternal (pulse rate, blood pressure, uterine contractions), as well as fetal (heart rate) monitoring will be performed every 15-30 minutes during the first 4 hours following the start of therapy then every 2 hours during the rest of treatment period. Patients whose contractions will stop after 48-72 hours will be observed for additional 24 hours to detect if contractions appear again so that if they remain stable, then they can be discharged and asked to come for follow-up after 1 week. As we stated in a previous work (13) that vaginal progesterone was effective for preventing recurrent PTL, thus all discharged patients will be advised to continue on progesterone till completed 36 weeks' gestation. In addition to progesterone treatment, all patients will be instructed to undergo periods of bed rest and, also they will be educated about the symptoms of PTL. The provided antenatal care will be at 2-weekly intervals till delivery. At any time if preterm contractions appeared re-admission with repeated treatment using the same drug will be used. At delivery, all data regarding the timing of labor onset, along with maternal and neonatal complications, will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients presented in outpatient clinic, admitted through emergency room or referred from any other hospitals will be the candidates for the study if they are of any age, any parity, carrying a singleton pregnancy, at a gestational age (GA) between 24 and 34 weeks, and whether or not they had a previous history of PTL.

Exclusion Criteria:

* The presence of major fetal anomaly, intrauterine fetal death, advanced cervical dilatation (>4cm), membranes bulging into the vagina in asymptomatic women, history of ruptured membranes, major antepartum hemorrhage, major chronic medical disorder (such as chronic hypertension, chronic renal disease, and pre-gestational diabetes mellitus as these conditions would increase the risk of PTL and potentially confound the primary study outcome), twins or higher order multiple pregnancy, any other condition in which continuation of the pregnancy can harm the mother or fetus and any contraindication for nifedipin and/or nicorandil therapy.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 227 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
the proportion of women remaining undelivered during the whole period of hospitalization. Treatment failure is considered in participants who delivered during this period, or those who need repeated treatment course. | 9 months

SECONDARY OUTCOMES:
readmission after discharge | 9 months
time (days) till delivery | 9 months
maternal outcomes (gestational age at delivery, mode of delivery, any complications during delivery) | 9 months
neonatal outcomes (weight, Apgar score, admission to neonatal intensive care unit | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: menoufia university, Study Chair — menoufia fuculty of medicine; Alhayah national hospital, Study Chair — Alhayah national hospital
Locations (2):
- Menoufia University, Shebin Elkom, Egypt
- Alhayah national hospital, Abhā, Saudi Arabia